CLINICAL TRIAL: NCT00818181
Title: A Multicentre Open Label Safety Study of a Sublingual Specific Immunotherapy With a Solution of Birch Pollen Allergen Extract in Patients With Clinically Relevant Birch Pollen Allergy
Brief Title: Open Label Safety Study of a Birch Pollen Allergen Extract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL0206st; 2007-006053-24 (EudraCT Number)
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Rhinoconjunctivitis
Keywords: Type I - Allergy, rhinoconjunctivitis

ARMS (1):
- Solution of birch pollen allergen extract (Experimental): In total up to 4 drops (dose for maintainace therapy)are administered under the tongue.
  Interventions: Drug: Biological: AL0206st

INTERVENTIONS:
Drug: Biological: AL0206st

SUMMARY:
This trial is performed to assess safety of a sublingual birch pollen extract.

ELIGIBILITY:
Inclusion Criteria:

* Allergic rhinoconjunctivitis attributable to birch pollen
* Positive SPT
* Positive EAST

Exclusion Criteria:

* Serious chronic diseases
* Other perennial allergies
* Partly controlled asthma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
number of patients with at least one adverse event | 8 months
  Between Visit 03 and Visit 05 (June 2008 - January 2009)

SECONDARY OUTCOMES:
Systemic reactions | Entire treatment period
  The occurrence of systemic reactions during the entire treatment period: For this purpose patients completed a diary covering the treatment phase.

OTHER OUTCOMES:
Immunologic parameters | during the course of the study
  Immunologic parameters (IgE, IgG1 and IgG4) were evaluated during the course of the study in order to obtain evidence of the immunologic effects.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Hunzelmann, Prof. Dr., Principal Investigator — University of Cologne
Locations (1):
- Prof. Dr. Nicolas Hunzelmann, Cologne, Germany

REFERENCES:
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de